CLINICAL TRIAL: NCT00373984
Title: A Study of the Incidence of Post-Thoracotomy Shoulder Pain
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Shoulderpain
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Post-thoracotomy Shoulder Pain
Keywords: shoulder; thoracotomy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Patients undergoing chest surgery (thoracotomy) often develop shoulder pain after their operation despite epidural pain control of the incision. We plan to study the incidence of this phenomenon in our institution to determine whether there are patterns that may predict those persons at highest risk of developing this type of pain. Further, we hope to determine whether newer surgical techniques have an impact on the development of this type of pain.

DETAILED DESCRIPTION:
Patients undergoing thoracic surgery often benefit from aggressive post-operative pain management including thoracic epidural analgesia (1). However, a significant number of patients develop shoulder tip pain (SP) refractory to epidural analgesia. The incidence of post-thoracotomy ISTP has been noted in association with treatment studies to be high, as much as 88% of patients having thoracotomy for lobectomy (2). The actual incidence of SP has not been systematically studied. We propose to prospectively study all thoracotomy patients for a period of six months. The goal of this study is to determine the incidence of post-thoracotomy SP and to identify predictive factors. Further, we hope to elucidate the incidence of SP associated with newer minimally invasive surgical procedures such as video-assisted thoracoscopic surgery for lobectomy. This will facilitate early identification of the patients most likely to benefit from treatment.

All procedures requiring thoracotomy including video assisted thoracoscopic surgery (VATS) be included. The following non-nominal information will be collected:1. demographic data- age, sex, BMI, 2. presence/absence and tip position of epidural catheter3. type of surgery and duration of surgery4. surgeon5. inta-operative analgesia6. epidural infusion and rate7. position and number of chest drains8. pain assessment9. co-morbid conditions- diabetes, hypertension, coronary artery disease, pulmonary disease (obstructive/restrictive), arthritis (rheumatoid/osteo)10. pre-existing pain conditions 11. treatment for ISTPPatients will be separated into two groups for assessment of SP. The two groups will consist of patients with functional epidural analgesia (group E) and those without epidural catheters or with non-functioning epidural catheters (group NE). Epidural catheter level will be determined using nerve stimulation (Tsui test) prior to induction of anesthesia. Upon arrival to the Post Anesthetic Care Unit (PACU), patients in group E will be assessed for incision pain and shoulder tip pain. Epidural catheter function will be assessed by pinprick testing to assess the function of the anesthetic. In patients experiencing incisional pain and in whom nerve stimulation indicates positioning of the epidural catheter in the epidural space (stimulation at 1.1-10 mA), 4 millilitres of 2% lidocaine will be infused through the epidural catheter. Incision pain and anesthetic level will be reassessed after 10 minutes. The catheter will be considered non-functional if no improvement in incisional pain is noted 10 minutes after infusion of the 2% lidocaine. Time 0 will be the time at which incisional pain is determined by pinprick testing to be absent. This may be immediately on arrival to PACU or 10 minutes after instillation of 2% lidocaine. Standard epidural infusions of bupivacaine 0.1% plus hydromorphone 0.015mg/ml or ropivacaine 0.1% will be continued. Management of SP will be at the discretion of the attending anesthesiologist and the Acute Pain Service. Patients will be followed daily until resolution of the SP or hospital discharge. Patients with ongoing ISTP at discharge will be followed by telephone weekly for 3 months or until the pain resolves, whichever is earlier. Patients in group NE will also be assessed for incision and shoulder tip pain upon arrival to the PACU. VAS and VRS will be obtained after the initial nursing assessment. This will be recorded as time 0. Patients will be asked to identify the area of greatest pain. They will then be asked specifically about shoulder tip pain. VRS and VAS scores will be recorded for 1) incision pain, 2) ipsilateral shoulder pain 3) contralateral shoulder pain and 4) area of greatest pain if different from 1,2and 3. Management of pain will be at the discretion of the anesthesiologist and the Acute Pain Service. Patients will be followed until the resolution of their pain or until discharge. Patients with ongoing SP at discharge will be followed by telephone weekly for three months or until the pain resolves, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* All procedures requiring thoracotomy including video assisted thoracoscopic surgery (VATS) be included.

Exclusion Criteria:

* Age less than 18 years
* Inability to communicate in English
* surgery in a position other than lateral ie. supine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Primary Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Slinger, MD, Principal Investigator — Anesthesiologist
Locations (1):
- Toronto General Hospital, 200 Elizabeth St., Toronto, Ontario, Canada